CLINICAL TRIAL: NCT03048591
Title: The Exploratory Study of Electroacupuncture in the Treatment of Peripheral Neuropathy Induced by Platinum Based Chemotherapy Drugs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: E2016014A
Record Dates: First submitted 2017-02-07; First posted 2017-02-09 (Estimated); Last update posted 2018-02-12 (Actual); Status verified 2017-02

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy
MeSH Terms: interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electroacupuncture group (Experimental)
  Interventions: Device: electroacupuncture
- control group (No Intervention)

INTERVENTIONS:
Device: electroacupuncture — Acupoint selection: Bilateral Hegu (LI4), Qu-chi (LI1) of upper limbs and bilateral Zusanli (ST36) ,Taichung (LR3)of lower limbs.
  Arms: Electroacupuncture group

SUMMARY:
Through the research to confirm the effectiveness and safety of using electroacupuncture in the treatment of chemotherapy-induced peripheral neuropathy.

ELIGIBILITY:
Inclusion Criteria:

1. The histopathological and / or cellular pathology results prove malignancy of the tumor and the patient has received chemotherapy treatment before.
2. 15weeks after the completion of chemotherapy, the limbs are still feeling abnormal and the symptoms fulfill World Health Organization (WHO) grade 2 or more.
3. zubrod - Eastern Cooperative Oncology Group-WHO (ZPS) grade 0-2, cardiac function, liver function and renal function are not significantly abnormal, the survival period of the patient is expected to be more than 6 months.
4. Gender unrestricted, aged between 18 to 80 years old.
5. Voluntary participation in the study, will to sign informed consent, willing to comply with randomized grouping, will to follow-up.

Exclusion Criteria:

1. Patients who suffer from peripheral neuropathy due to infection, radiotherapy, HIV, chronic alcoholism, hypothyroidism, diabetes, paraneoplastic syndrome or other diseases; or are suffering from nervous system diseases.
2. Patients who are being treated with other drugs that may lead to neurotoxicity .
3. Patients with blood coagulation disorder.
4. Pregnancy and lactating women.
5. Patients with infection, scarring or defects near the acupoint sites.
6. Received intervention for the prevention and treatment of peripheral neuropathy 2 weeks before screening or has received traditional Chinese medicine (acupuncture, moxibustion, cupping, Chinese medicine therapy one month before.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2018-02-10 (Estimated); Primary Completion 2018-09-01 (Estimated); Study Completion 2018-11-01 (Estimated)

PRIMARY OUTCOMES:
Quality of life questionnaire to assess chemotherapy-induced peripheral neuropathy (QLQ-CIPN20) | 6 weeks

SECONDARY OUTCOMES:
Functional Assessment of Cancer Treatment - General scale（FACT-G） | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bin Wang, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital